CLINICAL TRIAL: NCT02758457
Title: Zirconia-based and Metal-based Single Crown Posterior Restorations: 5-year Results of a Randomized Controlled Clinical Study.
Brief Title: Zirconia and Metal-based Single Crown Posterior Restorations.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, carlo monaco, Dr. Carlo Monaco, DDS, PhD, University of Bologna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 222893
Record Dates: First submitted 2016-04-23; First posted 2016-05-02 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Dental Crowns; Dental Prosthesis; Prosthodontics
Keywords: cad/cam; dental porcelain; zirconia; press on metal
MeSH Terms: interventions — Crowns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- metal-based restorations (Active Comparator): single crown with a metal framework and pressed ceramic
  Interventions: Device: dental crowns
- zirconia-based restorations (Experimental): single crown with a zirconia framework and pressed ceramic
  Interventions: Device: dental crowns

INTERVENTIONS:
Device: dental crowns

SUMMARY:
The objective of this study was to compare the 5-year survival and clinical behavior of single posterior ceramic crowns made with pressable ceramic on zirconia or on a metal framework. If failures occurred, the further aim of the study was to delineate the factors contributing to the failure. The null hypothesis stated that the survival of zirconia-based restorations would be no worse that those made with metal-based material.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Male and female patients from 18-70 years of age
* Need for a single crown restoration
* Presence of antagonist
* minimum of 20 teeth
* moderate to good oral hygiene with the ability to perform mechanical oral hygiene techniques including tooth brushing
* low to moderate caries risk, and no active periodontal disease.

Exclusion Criteria:

* Women who are pregnant at the date of inclusion
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Smoking more than 15 cigarettes a day
* Poor oral hygiene (Plaque Index over 30%)
* Bruxism
* vital teeth
* allergic reaction or hypersensitivity to ingredients of the adhesive or restorative material

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2008-01; Primary Completion 2013-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Technical complication rate | 5 years
  assessed by USPHS-criteria

SECONDARY OUTCOMES:
Survival rate | 1, 3, 5 years
  assessed by bleeding on probing
Survival rate | 1, 3, 5 years
  pocket probing depth

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical and Neuromotor Sciences, Division of Prosthotontics and Maxilla-Facial Rehabilitation, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Monaco C, Llukacej A, Baldissara P, Arena A, Scotti R. Zirconia-based versus metal-based single crowns veneered with overpressing ceramic for restoration of posterior endodontically treated teeth: 5-year results of a randomized controlled clinical study. J Dent. 2017 Oct;65:56-63. doi: 10.1016/j.jdent.2017.07.004. Epub 2017 Jul 21. PMID 28736293